CLINICAL TRIAL: NCT02748681
Title: Home Polygraphic Recording With Telemedicine Monitoring for Diagnosis and Treatment of Sleep Apnea in Stroke (HOPES)
Brief Title: Telemedicine Monitoring of Sleep Apnea in Stroke
Acronym: HOPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurologisches Rehabiliationszentrum Rosenhügel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOPESV3
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Stroke; Sleep Apnea
Keywords: obstructive sleep apnea; CPAP; stroke; telemedicine; neurorehabilitation; systolic blood pressure
MeSH Terms: conditions — Stroke; Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine Group (Active Comparator): Patient group with a telemedicine monitoring system
  Interventions: Device: Auto CPAP AirSense™ 10(Resmed)
- Standard Group (Active Comparator): Patient Group without a telemedicine monitoring
  Interventions: Device: Auto CPAP AirSense™ 10(Resmed)

INTERVENTIONS:
Device: Auto CPAP AirSense™ 10(Resmed) — AutoSet CPAP without telemedicine monitoring

SUMMARY:
Study Objectives:

Meta-analyses report a high prevalence of moderate to severe sleep apnea of more than 50% in stroke patients, with adherence rates for CPAP therapy of only 30%.

The primary objective of this study is to determine whether CPAP adherence in stroke patients with obstructive sleep apnea can be improved by a CPAP training strategy during rehabilitation combined with a telemedicine monitoring system after discharge.

The secondary objective is to compare recording quality as well as subjective and objective sleep data of non-attended level III polygraphy, polysomnography and telemetric CPAP data in the management of sleep apnea in stroke.

Further the investigators aim to study changes in nocturnal systolic blood pressure due to CPAP therapy with the pulse transit time method.

Finally, the investigators intend to study the relationship between CPAP compliance, sleep and medical and neurorehabilition outcome parameters.

Design:

Single-blind, mono-center, randomized controlled trial on standard CPAP treatment as compared with CPAP treatment with a telemedicine monitoring system in stroke patients with moderate to severe OSA.

Setting: Neurorehabilitation center in Vienna, Austria

Patients: Adult subacute (1 to 12 months post stroke) stroke patients 18-70 yrs of age) with moderate to severe OSA (apnea hypopnea index (AHI) ≥ 15/hr) determined by non-attended polysomnography (AHI) ≥ 15/hr of sleep) or level III polygraphy (AHI) ≥ 30/hr of out-of-center sleep testing (OCST), who undergo successful CPAP training and titration (goal AHI< 10) at the neurorehabilitation unit.

Interventions: Patients will be randomized to either standard care with an autotitrating CPAP device or an autotitrating CPAP device that transmits physiologic information (i.e., adherence, air leak, residual AHI) daily to a website that will be reviewed by their homecare provider. If any problems are identified, the patient will be contacted by his homecare provider by telephone. Neurologists performing sleep and neurological scoring will be blinded to the randomization.

Measurements: Recording of the different measuring systems, subjective and objective sleep quality, CPAP adherence after 3 months and 1 year in hours used per night, systolic BP determined by means of a non-linear algorithm and an individual one-point calibration of the pulse transit time obtained with a cuff-based BP measuring system (SOMNOmedics GmbH, Germany) and neurorehabilitation outcome parameters as Barthel Index, Timed Up and Go Test.

DETAILED DESCRIPTION:
The investigators intend to perform a single-blind, mono-center, randomized controlled trial on standard CPAP treatment as compared with CPAP treatment with a telemedicine monitoring system in stroke patients with moderate to severe OSA.

Patients accepting CPAP therapy after successful titration will be randomized to either a standard care or a telemedicine group (1:1 ratio) and will subsequently be informed about the study arm by their homecare provider. The study was approved by the Clinical Research Ethics Board of the public health services of Vienna.

Written informed consent for all examinations will be obtained upon patients' admission. If patients agree to undergo CPAP monitoring, further informed consent will be obtained. The study will be performed in accordance with the relevant guidelines of the Declaration of Helsinki, 1964, as amended in Tokyo, 1975, Venice, 1983, Hong Kong, 1989, and Somerset West, 1996.

Screening Sleep Studies

Over the four to eight weeks of neurorehabilitation, each stroke patient ( 19-70 yrs of age) will be offered a nocturnal respirographic screening evaluation of SA (see study flow chart). Within the study period the investigators expect to screen 170 patients per year.

Diagnosis of sleep apnea and referral to CPAP training:

SA and referral to CPAP training will be based on an AHI ≥ 15/h sleep, as recommended by an international task force on the standardization of definitions for sleep-related breathing disorders to indicate moderate SA .

If screening with type-3 polygraphy reveals an AHI ≥ 15 and ≤ 30/h of recording time or if subjective sleep time in the concomitant sleep log is less than 4 hours, non-attended polysomnography will be performed to confirm the diagnosis of SA. If type-3 polygraphy shows an AHI of ≥ 30/h recording time, the patient will directly be referred to CPAP therapy.

Polysomnography and polygraphy will be performed by a trained staff member using the Somnomedics Diagnostic Systems (SOMNOmedics GmbH, Germany). Patients will be studied in their hospital beds. Polygraphic and polysomnographic all-night recordings according to AASM standard criteria will be obtained between approximately 22.00 (lights-out) and 6.00 am (buzzer or alarm clock). Thus, time in bed (TIB) is fixed with 7.5 hours.

Polygraphic recording includes nasal air flow, snore train, thoracic and abdominal effort, oxyhemoglobin saturation, and determination of the body position. Recordings will be used in further investigations if at least 4 h of data can be obtained. EEG sleep data will include 6 EEG channels (F3-A2, F4-A1, C3-A2, C4-A1, O1-A2, O2-A1) according to the 10/20 system, 2 electrooculogram (EOG) channels (left/right), submental electromyogram (EMG) and tibialis anterior electromyogram from both legs (EMG) and will be scored manually.

Systolic BP will be determined by means of a non-linear algorithm and an individual one-point calibration of the pulse transit time obtained with a cuff-based BP measuring device (SOMNOmedics GmbH, Germany). The number of systolic rises (defined as >15mmHg) in relation to respiratory events and the maximum systolic blood pressure will be determined.

Patients will be asked to complete the Self-Assessment Scale for Sleep and Awakening Quality (SSA) according to Saletu et al. (1987).

Polygraphic data recordings will be manually scored for apneas and hypopneas according to the criteria developed by the American Academy of Sleep Medicine (AASM). For scoring an event as a hypopnea, a 30% reduction of nasal flow associated with an oxygen desaturation of at least 3% is required. The AHI is defined as the sum of all apneas and hypopneas occurring per hour of recording time.

CPAP Protocol

All patients referred to CPAP therapy will receive a 60-min PAP training. A nasal or oronasal mask will be fitted to the patient's face by the PAP coordinator of our center, who is a trained respiratory therapist and ESRS-certified somnologist (MS) with many years of experience in sleep apnea patients.

Patients will be provided with an AirSense™ 10 AutoSet CPAP (Resmed) including a humifdifier. This auto-titrating device monitors patients' airflow and adjusts pressure automatically to eliminate sleep apnea.

The AirSense 10 AutoSet is able to differentiate between obstructive and central apneas. It is set to auto-titrate at pressures between 6 and 13 cm H2O, which reflects our current clinical practice. Pressure limits can be increased up to 16 cm H2O, but will be decreased to the smallest range leading to a normalized AHI in order to avoid overtitration.

Patients accepting CPAP therapy after the training session will be motivated to use it for at least 4 > hours sleep/night over one week. Additional nocturnal pulse oximetry will be obtained. Patients will be coached by trained nurses during the night. Relatives will also be trained in using the humidifier and cleaning the mask and the humidifier chamber. Data card AHI, oximetry and leakage information will be collected every day. Pressure limits can be increased or decreased to improve patient comfort. If patients consider the interface uncomfortable, it may be changed.

After one week, patients with a median CPAP use of >4/hours will undergo unattended CPAP polysomnography.

The quality of CPAP titration is graded as follows: optimal (obstructive AHI ≤ 5/h, supine REM sleep on the treatment pressure; desaturation index≤ 5/h of sleep), good (obstructive AHI < 10/h, REM sleep on the treatment pressure, desaturation index≤ 10/h), adequate (AHI < 10/h, supine NREM sleep on the treatment pressure, desaturation index≤ 10/h). A persisting central AHI < 5 will be tolerated. If none of these criteria are met, patients will be referred to conventional attended CPAP polysomnograpy and excluded from the study.

Patients who chose to participate in the telemetric study part will be asked to sign informed consent and will be randomized to either a standard care or a telemedicine group (1:1 ratio) using sequentially numbered envelopes prepared by the CPAP homecare provider.

After receiving their prescribed CPAP device by their homecare provider they will be informed in which group they are.

Study staff performing sleep recordings and clinical ratings will be blinded to the study arm. In case of treatment pressure changes doctors will be informed about the study arm.

Clinical Scales

In both study arms patients will be asked to complete the following scales:

ESS (Epworth Sleepiness Scale) SSA (Self-Assessment Scale for Sleep and Awakening Quality according to Saletu et al. 1987) QoL (Quality of Life Index according to Mezzich et al.) BQ (Berlin Questionnaire) PAP Satisfaction Questionnaire

NIH Stroke Scale (National Institute of Health, National Institute of Neurological Disorders and Stroke) TUG (Timed Up and Go Test) NHPT (Nine Hole Peg Test) BI (Barthel Index) Moca Test

Outpatient Monitoring after Randomization

Standard Care

Patients will be contacted by their homecare provider 2 days after receiving their CPAP device and will be asked about progress and adherence,as well as about any problems that might have occurred. After 3 months of therapy, patients will return to the hospital to see the PAP coordinator and their doctor. Data on a variety of physiological variables, including PAP adherence, PAP pressure applied, mask leakage, and residual respiratory events, will be downloaded from their CPAP devices. Any problems with treatment may be addressed.

Patients will be asked to complete a number of clinical scales and answer a variety of survey questions concerning side effects and sleep quality.

A non-attended PSG will be performed at the patients' homes.

Telemedicine Like in standard care, patients will receive an AirSense™ 10 AutoSet CPAP. In addition, the telemedicine module of the PAP device will be activated by the homecare provider. The module will be programmed to send physiological information (PAP adherence, PAP pressure applied, mask leakage and residual respiratory events) to a web-based database via a GPRS module every day.

Patients will be contacted by the homecare provider after 2 days and will be asked about progress and compliance as well as about any problems. The PAP coordinator at the homecare provider will review the downloaded information every morning except on weekends and holidays and will contact the patient if any of the following occur: mask leakage of the 95 percentile > 24 L/min, < 4 h of use for two consecutive nights, AHI > 10 events/h, and 90th percentile of pressure > 16 cm H2O. The homecare provider will call the patient or his/her relatives and will ask about symptoms such as dry mouth, mask issues, discomfort with the device, or any other problems. If the only issue is low adherence due to lack of motivation, the homecare provider will encourage the patient to use PAP. Should there be any other problems, the homecare provider will discuss the case with the PAP coordinator (the same person that sees the patients in the standard arm) and arrange for the patient to talk to or see the PAP coordinator, depending on the patient's responses and the physiological data obtained. Specific interventions may be performed to improve compliance that are considered standard at the hospital (e.g., different mask, chin strap, modifications of pressure settings, modifications of humidifier settings, saline nasal sprays).

After 3 months of therapy, patients will return to the hospital to see their doctor and the data obtained will be reviewed (including CPAP pressure, mask leakage, residual respiratory events, and compliance). Any problems with treatment may be addressed.

Like in the standard arm, polysomography will be performed at the patients' homes and clinical scales will be completed.

Time Spent with Patients

The time our research coordinator or PAP coordinator spends with patients will be recorded and written in a daily log sheet. This includes time spent fitting masks, problem solving, talking with patients on the phone, meeting with patients, and reviewing downloaded or transmitted information.

Statistical Analyses

Statistical analyses will be performed in SPSS version 10 for Windows (SPSS Inc. Chicago, IL, USA). All P-values are two-sided and values < 0.05 are considered statistically significant. To examine and compare demographic and test characteristics at inclusion, chi-sqare test, t-test and Mann-Whitney U-test for independent samples will be used according to distribution, which will be examined with the Kolmogorov-Smirnov Test. The primary outcome is PAP adherence after 3 months (min used per day). To calculate the number of participants needed for an effect size larger than 0,80 as proposed by Cohen (Statistical power analysis for behavioural science. 1988), the investigators based a power calculation on the results of the study by Fox et al. in patients with sleep apnea, comparing telemedicine versus standard CPAP treatment over 3 months. The result of this calculation was 11 patients in one group. Considering patients who will discontinue CPAP treatment, the investigators aim to include 55 patients in the randomisation process. Based on previous data the investigators consider that 168 patients will have to be included in the screening process for sleep apnea.

Clinical variables will be correlated with compliance data. Therefore the spearman rank correlation coefficient and the pearson correlation coefficient will be used. Blood pressure data at baseline and after 3 months of CPAP treatment will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-70 yrs of age) with a subacute stroke (1-12 months)
* Diagnosis of sleep apnea and acceptance of CPAP therapy:

Exclusion Criteria:

* Patients with sopor/coma
* Any form of dementia (Mini-Mental State Examination <20)
* Previously diagnosed sleep apnea and established CPAP therapy
* Purely central sleep apnea
* Chronic obstructive pulmonary disease more than Gold III
* Cancer
* Severe kidney diseases
* Coexisting causes of daytime sleepiness (e.g. narcolepsy, night or rotating shift-work; self-reported average sleep duration <4 h)
* A major psychiatric or any other acute medical condition
* Patients unable or unwilling to comply with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
CPAP adherence in minutes used per night | after 3 months

SECONDARY OUTCOMES:
systolic BP | Change from baseline systolic blood pressure to CPAP systolic blood pressure at three months

OTHER OUTCOMES:
Barthel Index | Change from baseline score to score under CPAP therapy at three months

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Saletu, MD, Study Director — Neurological Rehabilitation Center Rosenhügel Rosenhügelstrasse 192a, A-1130
Locations (1):
- Michael Saletu, MD, Vienna, Austria

REFERENCES:
- [Derived] Kotzian ST, Saletu MT, Schwarzinger A, Haider S, Spatt J, Kranz G, Saletu B. Proactive telemedicine monitoring of sleep apnea treatment improves adherence in people with stroke- a randomized controlled trial (HOPES study). Sleep Med. 2019 Dec;64:48-55. doi: 10.1016/j.sleep.2019.06.004. Epub 2019 Jun 13. PMID 31670004
- [Derived] Saletu MT, Kotzian ST, Schwarzinger A, Haider S, Spatt J, Saletu B. Home Sleep Apnea Testing is a Feasible and Accurate Method to Diagnose Obstructive Sleep Apnea in Stroke Patients During In-Hospital Rehabilitation. J Clin Sleep Med. 2018 Sep 15;14(9):1495-1501. doi: 10.5664/jcsm.7322. PMID 30176970
- [Derived] Kotzian ST, Schwarzinger A, Haider S, Saletu B, Spatt J, Saletu MT. Home polygraphic recording with telemedicine monitoring for diagnosis and treatment of sleep apnoea in stroke (HOPES Study): study protocol for a single-blind, randomised controlled trial. BMJ Open. 2018 Jan 9;8(1):e018847. doi: 10.1136/bmjopen-2017-018847. PMID 29317418